CLINICAL TRIAL: NCT04659161
Title: A Phase 3, Randomized, Double-blind, Parallel-group, Placebo-controlled, Multicenter Study to Evaluate the Efficacy and Safety of KarXT in Acutely Psychotic Hospitalized Adults With DSM-5 Schizophrenia
Brief Title: A Study to Assess Efficacy and Safety of KarXT in Acutely Psychotic Hospitalized Adult Patients With Schizophrenia (EMERGENT-2)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KAR-007
Record Dates: First submitted 2020-12-02; First posted 2020-12-09 (Actual); Results first posted 2023-12-12 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Schizophrenia; Schizophrenia; Psychosis
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders | interventions — xanomeline; trospium chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- KarXT (Experimental)
  Interventions: Drug: Xanomeline and Trospium Chloride Capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xanomeline and Trospium Chloride Capsules — Oral xanomeline 50 mg/trospium chloride 20 mg BID (twice a day) for the first 2 days (Days 1 and 2) followed by xanomeline 100 mg/trospium chloride 20 mg BID for the remainder of Week 1 (Days 3 to 7). At Visit 5 (Day 8), dosing was to be titrated upwards to xanomeline 125 mg/trospium chloride 30 mg BID unless the subject was continuing to experience adverse events (AEs) from the previous dose of KarXT 100/20 BID. All subjects who were increased to KarXT 125/30 BID, depending on clinical response and tolerability, had the option to return to KarXT 100/20 BID for the remainder of the treatment period.
  Other Names: KarXT
  Arms: KarXT
Drug: Placebo — Placebo Capsules twice a day (BID)
  Other Names: PBO
  Arms: Placebo

SUMMARY:
This is a Phase 3, randomized, double-blind, parallel-group, placebo-controlled, multicenter inpatient study to examine the efficacy and safety of KarXT in adult subjects who are acutely psychotic with a Diagnostic and Statistical Manual Fifth Edition (DSM-5) diagnosis of schizophrenia. The primary objective of the study is to assess the efficacy of KarXT (a fixed combination of xanomeline 125 mg and trospium chloride 30 mg twice daily [BID]) versus placebo in reducing Positive and Negative Syndrome Scale (PANSS) total scores in adult inpatients with a DSM-5 diagnosis of schizophrenia. The secondary objectives of the study are to evaluate improvement in disease severity and symptoms, safety and tolerability, and pharmacokinetics in adult inpatients with a DSM-5 diagnosis of schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is aged 18 to 65 years, inclusive, at screening.
2. Subject is capable of providing informed consent.

   1. A signed informed consent form must be provided before any study assessments are performed.
   2. Subject must be fluent (oral and written) in English to consent
3. Subject has a primary diagnosis of schizophrenia established by a comprehensive psychiatric evaluation based on the DSM-5 criteria and confirmed by Mini International Neuropsychiatric Interview for Schizophrenia and Psychotic Disorder Studies (MINI) version 7.0.2.
4. Subject is experiencing an acute exacerbation or relapse of psychotic symptoms, with onset less than 2 months before screening.

   1. The subject requires hospitalization for this acute exacerbation or relapse of psychotic symptoms.
   2. If already an inpatient at screening, has been hospitalized for less than 2 weeks for the current exacerbation at the time of screening.
5. Positive and Negative Syndrome Scale total score between 80 and 120, inclusive. Score of ≥4 (moderate or greater) for ≥2 of the following Positive Scale (P) items:

   1. Item 1 (P1; delusions)
   2. Item 2 (P2; conceptual disorganization)
   3. Item 3 (P3; hallucinatory behavior)
   4. Item 6 (P6; suspiciousness/persecution)
6. Subjects with no change (improvement) in PANSS total score between screening and baseline (Day -1) of more than 20%.
7. Subject has a CGI-S score of ≥4 at screening and baseline (Day -1) visits.
8. Subject will have been off lithium therapy for at least 2 weeks before baseline and free of all oral antipsychotic medications for at least 5 half-lives or 1 week, whichever is longer, before baseline (Day -1).
9. Subjects taking a long-acting injectable antipsychotic could not have received a dose of medication for at least 12 weeks (24 weeks for INVEGA TRINZA) before baseline visit (Day -1).
10. Subject is willing and able to be confined to an inpatient setting for the study duration, follow instructions, and comply with the protocol requirements.
11. BMI must be ≥18 and ≤40 kg/m2.
12. Subject resides in a stable living situation and is anticipated to return to that same stable living situation after discharge, in the opinion of the investigator.
13. Subject has an identified reliable informant.
14. Women of childbearing potential, or men with sexual partners of childbearing potential, must be able and willing to use at least 1 highly effective method of contraception during the study and for 30 days after the last dose of study drug. Sperm donation is not allowed for 30 days after the final dose of study drug.

Exclusion Criteria:

1. Any primary DSM-5 disorder other than schizophrenia within 12 months before screening (confirmed using MINI version 7.0.2 at screening). Symptoms of mild mood dysphoria or anxiety are allowed as long as these symptoms are not the primary focus of treatment. A screening subject with mild substance abuse disorder within the 12 months before screening must be discussed and agreed upon with the medical monitor before they can be allowed into the study.
2. Subjects who are newly diagnosed or are experiencing their first treated episode of schizophrenia.
3. History or presence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic, or oncologic disease or any other condition that, in the opinion of the investigator, would jeopardize the safety of the subject or the validity of the study results.
4. Subjects with HIV, cirrhosis, biliary duct abnormalities, hepatobiliary carcinoma, and/or active hepatic viral infections based on either medical history or liver function test results.
5. History or high risk of urinary retention, gastric retention, or narrow-angle glaucoma.
6. History of irritable bowel syndrome (with or without constipation) or serious constipation requiring treatment within the last 6 months.
7. Risk for suicidal behavior during the study as determined by the investigator's clinical assessment and Columbia-Suicide Severity Rating Scale (C-SSRS).
8. Clinically significant abnormal finding on the physical examination, medical history, ECG, or clinical laboratory results at screening.
9. Subjects cannot currently (within 5 half-lives or 1 week, whichever is longer, before baseline [Day -1]) be receiving oral antipsychotic medications; monoamine oxidase inhibitors; anticonvulsants (eg, lamotrigine, Depakote); tricyclic antidepressants (eg, imipramine, desipramine); selective serotonin reuptake inhibitors; or any other psychoactive medications except for as needed anxiolytics (eg, lorazepam, chloral hydrate).
10. Pregnant, lactating, or less than 3 months postpartum.
11. If, in the opinion of the investigator (and/or Sponsor), subject is unsuitable for enrollment in the study or subject has any finding that, in the view of the investigator (and/or Sponsor), may compromise the safety of the subject or affect his/her ability to adhere to the protocol visit schedule or fulfill visit requirements.
12. Positive test for coronavirus (COVID-19) within 2 weeks before screening and at screening.
13. Subjects with extreme concerns relating to global pandemics, such as COVID-19, that preclude study participation.
14. Subject has had psychiatric hospitalization(s) for more than 30 days (cumulative) during the 90 days before screening.
15. Subject has a history of treatment resistance to schizophrenia medications defined as failure to respond to 2 adequate courses of pharmacotherapy (a minimum of 4 weeks at an adequate dose per the label) or required clozapine within the last 12 months.
16. Subjects with prior exposure to KarXT.
17. Subjects who experienced any adverse effects due to xanomeline or trospium.
18. Participation in another clinical study in which the subject received an experimental or investigational drug agent within 3 months before screening.
19. Risk of violent or destructive behavior.
20. Current involuntary hospitalization or incarceration.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2020-12-16 (Actual); Primary Completion 2022-05-24 (Actual); Study Completion 2022-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Inder Kaul, MD, Study Director — Karuna Therapeutics
Locations (22):
- United States (22):
  - Woodland International Research Group, LLC, Little Rock, Arkansas
  - CITrials, Bellflower, California
  - ProScience Research Institute, Culver City, California
  - California Clinical Trials Medical Group, Glendale, California
  - Synergy San Diego, Lemon Grove, California
  - CNS Network, Long Beach, California
  - Catalina Research Institute, LLC, Montclair, California
  - NRC Research Institute, Orange, California
  - California Neuropsychopharmacology Clinical Research Institute, Pico Rivera, California
  - California Neuropsychopharmacology Clinical Research Institute, San Diego, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Innovative Clinical Research, Inc., Miami Lakes, Florida
  - Research Centers of America, Oakland Park, Florida
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Pillar Clinical Research, Lincolnwood, Illinois
  - Arch Clinical Trials, St Louis, Missouri
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, Marlton, New Jersey
  - Neuro-Behavioral Clinical Research, North Canton, Ohio
  - Community Clinical Research, Austin, Texas
  - Pillar Clinical Research, Richardson, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yeung PP, Breier A, Zhu H, Kaul I, Marcus RN. Xanomeline and Trospium Chloride for the Treatment of Agitation Associated With Schizophrenia: PANSS-Excited Component Results From 3 Randomized, Double-Blind, Placebo-Controlled EMERGENT Trials. J Clin Psychiatry. 2025 Mar 24;86(2):24m15668. doi: 10.4088/JCP.24m15668. PMID 40215379
- [Derived] Citrome L, Neugebauer NM, Meli AA, Kando J. Xanomeline and Trospium Chloride Versus Placebo for the Treatment of Schizophrenia: A Post Hoc Analysis of Number Needed to Treat, Number Needed to Harm, and Likelihood to Be Helped or Harmed. Neuropsychiatr Dis Treat. 2025 Apr 5;21:761-773. doi: 10.2147/NDT.S503494. eCollection 2025. PMID 40212458
- [Derived] Kaul I, Claxton A, Sawchak S, Sauder C, Brannan SK, Raj E, Ruan S, Konis G, Brown D, Cutler AJ, Marcus R. Safety and Tolerability of Xanomeline and Trospium Chloride in Schizophrenia: Pooled Results From the 5-Week, Randomized, Double-Blind, Placebo-Controlled EMERGENT Trials. J Clin Psychiatry. 2025 Feb 26;86(1):24m15497. doi: 10.4088/JCP.24m15497. PMID 40047530
- [Derived] Kaul I, Sawchak S, Correll CU, Kakar R, Breier A, Zhu H, Miller AC, Paul SM, Brannan SK. Efficacy and safety of the muscarinic receptor agonist KarXT (xanomeline-trospium) in schizophrenia (EMERGENT-2) in the USA: results from a randomised, double-blind, placebo-controlled, flexible-dose phase 3 trial. Lancet. 2024 Jan 13;403(10422):160-170. doi: 10.1016/S0140-6736(23)02190-6. Epub 2023 Dec 14. PMID 38104575

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 21 study centers in the United States.
Pre-assignment Details: A total of 407 participants were screened, 252 were randomized, and 251 participants were treated.
Groups:
- KarXT: Participants received oral capsule KarXT (xanomeline/trospium chloride BID) in a treatment period of 5 weeks. Participants were started on a lead in dose of xanomeline 50 mg/trospium chloride 20 mg twice a day (BID) for the first 2 days followed by xanomeline 100 mg/trospium chloride 20 mg BID for the remainder of Week 1 (Days 3 to 7). On Day 8, dosing was titrated upwards to xanomeline 125 mg/trospium chloride 30 mg BID unless the Participant was continuing to experience adverse events from the previous dose increase of xanomeline 100 mg/trospium chloride 20 mg BID. All Participants who were increased to xanomeline 125 mg/trospium chloride 30 mg BID, depending on clinical response and tolerability, had the option to return to xanomeline 100 mg/trospium chloride 20 mg BID for the remainder of the treatment period.
- Placebo: Participants received the matching placebo to KarXT orally twice daily for a treatment period of 5 weeks.
Period: Overall Study
Arm/Group | KarXT | Placebo
Started | 126 | 126
Completed | 94 | 100
Not Completed | 32 | 26
Not completed — Adverse Event | 10 | 6
Not completed — Withdrawal by Subject | 13 | 12
Not completed — Other | 9 | 8

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) population included all participants who were randomized to the study. Participants were analyzed according to randomized treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | KarXT | Placebo | Total
Number analyzed (Participants) | 126 | 126 | 252
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.6 (10.42) | 46.2 (10.78) | 45.9 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 95 | 95 | 190
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 11 | 25
  Not Hispanic or Latino | 111 | 114 | 225
  Unknown or Not Reported | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 97 | 92 | 189
  White | 26 | 31 | 57
  Asian | 2 | 1 | 3
  Other | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  United States | 126 | 126 | 252
Baseline PANSS Total Score [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of participants with schizophrenia. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale. It takes approximately 45 to 50 minutes to administer. The total score is the sum of all scales with a minimum score of 30 and a maximum score of 210. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms. Population: Measure Analysis Population Description: A total of 252 subjects were randomized (126 subjects in each group) at 21 sites, and a total of 251 subjects were treated (126 [100.0%] in the KarXT group and 125 [99.2%] in the placebo group) during the study.
  units on a scale
    number analyzed (Participants) | 126 | 125 | 251
    (all) | 98.3 (8.93) | 97.9 (9.71) | 98.1 (9.31)
Baseline PANSS Positive Score [Mean (Standard Deviation); unit: units on a scale] — Population: Measure Analysis Population Description: A total of 252 subjects were randomized (126 subjects in each group) at 21 sites, and a total of 251 subjects were treated (126 [100.0%] in the KarXT group and 125 [99.2%] in the placebo group) during the study.
  units on a scale
    number analyzed (Participants) | 126 | 125 | 251
    (all) | 26.8 (3.74) | 26.7 (3.97) | 26.7 (3.85)
Baseline PANSS Negative Score [Mean (Standard Deviation); unit: units on a scale] — Population: Measure Analysis Population Description: A total of 252 subjects were randomized (126 subjects in each group) at 21 sites, and a total of 251 subjects were treated (126 [100.0%] in the KarXT group and 125 [99.2%] in the placebo group) during the study.
  units on a scale
    number analyzed (Participants) | 126 | 125 | 251
    (all) | 22.9 (4.00) | 22.9 (3.82) | 22.9 (3.90)
Baseline PANSS General Psychopathology Score [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Syndrome Scale (PANSS) is a medical scale used for measuring symptom severity of participants with schizophrenia. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale. It takes approximately 45 to 50 minutes to administer. The total score is the sum of all scales with a minimum score of 30 and a maximum score of 210. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms. Population: Measure Analysis Population Description: A total of 252 subjects were randomized (126 subjects in each group) at 21 sites, and a total of 251 subjects were treated (126 [100.0%] in the KarXT group and 125 [99.2%] in the placebo group) during the study.
  units on a scale
    number analyzed (Participants) | 126 | 125 | 251
    (all) | 48.6 (5.79) | 48.4 (5.99) | 48.5 (5.88)
Baseline PANSS Marder Factor Negative Score [Mean (Standard Deviation); unit: units on a scale] — The Marder Factor Negative Score is derived from the Positive and Negative Syndrome Scale (PANSS) and consists of the sum of 5 negative scales (N) and 2 general scales (G) (N1. Blunted affect; N2. Emotional withdrawal; N3. Poor rapport; N4. Passive/apathetic social withdrawal; N6. Lack of spontaneity; G7. Motor retardation; and G16. Active social avoidance), with a minimum score of 7 and a maximum score of 49. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms. Population: Measure Analysis Population Description: A total of 252 subjects were randomized (126 subjects in each group) at 21 sites, and a total of 251 subjects were treated (126 [100.0%] in the KarXT group and 125 [99.2%] in the placebo group) during the study.
  units on a scale
    number analyzed (Participants) | 126 | 125 | 251
    (all) | 22.9 (4.97) | 22.5 (4.73) | 22.7 (4.85)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Total Score at Week 5
Description: The PANSS is a medical scale used for measuring symptom severity of participants with schizophrenia. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale. It takes approximately 45 to 50 minutes to administer. The total score is the sum of all scales with a minimum score of 30 and a maximum score of 210. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms.
Time Frame: Baseline and Week 5
Population: The Modified Intent-to-Treat (MITT) population included all participants who were randomized, received at least one dose of study medication, and had a baseline and at least one post-baseline PANSS assessment. Here, the number of participants analyzed indicates participants who were evaluable for this measure at given time points for each group.
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 117 | 119
score on a scale | -21.2 (1.652) | -11.6 (1.600)
Statistical Analysis 1: Comparison: KarXT vs Placebo; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures; LS mean difference = -9.6, 95% CI 2-sided [-13.9 to -5.2]; Statistics are from a mixed model for repeated measures (MMRM). The model includes the treatment group (KarXT or placebo), visit, and the interaction between the treatment group and visit as fixed factors, and baseline PANSS total score, site, age, and gender as covariates. An unstructured covariance matrix is used to model the correlation among repeated measurements and the denominator degrees of freedom are computed using the Kenward-Roger method

2. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Positive Score at Week 5
Description: The PANSS is a medical scale used for measuring symptom severity of participants with schizophrenia. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale. For positive symptoms in schizophrenia, participants are rated from 1 to 7 on each symptom scale, with a minimum score of 7 and a maximum score of 49. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms.
Time Frame: Baseline and Week 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 117 | 119
score on a scale | -6.8 (0.526) | -3.9 (0.512)
Statistical Analysis 1: Comparison: KarXT vs Placebo; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures

3. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Negative Score at Week 5
Description: The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. For negative symptoms in schizophrenia, participants are rated from 1 to 7 on each symptom scale, with a minimum score of 7 and a maximum score of 49. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms.
Time Frame: Baseline and Week 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Deviation); unit: score on a scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 117 | 119
score on a scale | -3.4 (0.479) | -1.6 (0.466)
Statistical Analysis 1: Comparison: KarXT vs Placebo; Test type: Superiority; p = 0.0055, Mixed Model Repeated Measures

4. Secondary Outcome: Change From Baseline in Positive and Negative Syndrome Scale (PANSS) Marder Factor Negative Score
Description: The Marder Factor Negative Score is derived from the Positive and Negative Syndrome Scale (PANSS) and consists of the sum of 5 negative scales (N) and 2 general scales (G) (N1. Blunted affect; N2. Emotional withdrawal; N3. Poor rapport; N4. Passive/apathetic social withdrawal; N6. Lack of spontaneity; G7. Motor retardation; and G16. Active social avoidance), with a minimum score of 7 and a maximum score of 49. A decrease in PANSS total score correlates with an improvement in schizophrenia symptoms.
Time Frame: Baseline and Week 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 117 | 119
score on a scale | -4.2 (0.530) | -2.0 (0.517)
Statistical Analysis 1: Comparison: KarXT vs Placebo; Test type: Superiority; p = 0.0022, Mixed Model for Repeated Measures

5. Secondary Outcome: Change From Baseline Clinical Global Impression - Severity (CGI-S) Score at Week 5
Description: The CGI-S modified asked the clinician 1 question: "Considering your total clinical experience, how mentally ill is the participant at this time?" The clinician's answer rated on the following 7-point scale: 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants.
Time Frame: Baseline and Week 5
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 117 | 119
score on a scale | -1.2 (0.103) | -0.7 (0.099)
Statistical Analysis 1: Comparison: KarXT vs Placebo; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures

6. Secondary Outcome: Percentage of Positive and Negative Syndrome Scale (PANSS) Responders (>=30% Change in PANSS Total Score) at Week 5
Description: The PANSS is a medical scale used for measuring symptom severity of participants with schizophrenia. The PANSS rating form contains 7 positive symptom scales, 7 negative system scales, and 16 general psychopathology symptom scales. Participants are rated from 1 to 7 on each symptom scale. The total score is the sum of all scales with a minimum score of 30 and a maximum score of 210. A PANSS responder is defined as a participant with at least a 30% change in PANSS total score compared to baseline at Week 5.
Time Frame: Baseline and Week 5
Population: The Modified Intent-to-Treat (MITT) population included all participants who were randomized, received at least one dose of study medication, and had a baseline and at least one post-baseline PANSS assessment. Here, the number of participants analyzed indicates participants who were evaluable for this measure at given time points for each group. The overall number of participants was analyzed (N) = number of subjects with Week 5 score.
Measure: Count of Participants; unit: Participants
Arm/Group | KarXT | Placebo
Number analyzed (Participants) | 93 | 99
Participants | 51 | 28
Statistical Analysis 1: Comparison: KarXT vs Placebo; Test type: Superiority; p < 0.0001, Mixed Model for Repeated Measures

ADVERSE EVENTS:
Time Frame: From the start of study drug administration up to Week 5.
Description: The Safety population included all participants who received at least one dose of study medication.
Arm/Group | KarXT | Placebo
All-Cause Mortality (participants affected / at risk) | 0/126 | 0/125
Serious Adverse Events (participants affected / at risk) | 2/126 | 2/125
Other Adverse Events (participants affected / at risk) | 95/126 | 73/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | KarXT (N=126) | Placebo (N=125)
Appendicitis (Infections and infestations) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 0 — Suicidal ideation
Schizophrenia (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | KarXT (N=126) | Placebo (N=125)
Constipation (Gastrointestinal disorders) | 27 | 13
Dyspepsia (Gastrointestinal disorders) | 24 | 10
Nausea (Gastrointestinal disorders) | 24 | 7
Vomiting (Gastrointestinal disorders) | 18 | 1
Abdominal discomfort (Gastrointestinal disorders) | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 4
Dry mouth (Gastrointestinal disorders) | 6 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 2
Toothache (Gastrointestinal disorders) | 1 | 5
Headache (Nervous system disorders) | 17 | 15
Dizziness (Nervous system disorders) | 11 | 4
Somnolence (Nervous system disorders) | 6 | 5
Anxiety (Psychiatric disorders) | 6 | 5
Agitation (Psychiatric disorders) | 2 | 8
Insomnia (Psychiatric disorders) | 3 | 6
Psychotic disorder (Psychiatric disorders) | 1 | 6
Hypertension (Vascular disorders) | 12 | 1
Orthostatic hypotension (Vascular disorders) | 3 | 1
Heart rate increased (Investigations) | 4 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 3
Vision blurred (Eye disorders) | 6 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 3 | 0
Tachycardia (Cardiac disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2021-08-09): https://cdn.clinicaltrials.gov/large-docs/61/NCT04659161/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-28): https://cdn.clinicaltrials.gov/large-docs/61/NCT04659161/SAP_001.pdf